CLINICAL TRIAL: NCT06146205
Title: The Hip Fracture Surgical Approach Trial
Acronym: HIFSAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Oslo University Hospital (Other); University Hospital, Akershus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HIFSAT
Record Dates: First submitted 2023-11-08; First posted 2023-11-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hip Fracture; Femoral Neck Fracture
Keywords: Fragility fracture; Surgical approach; Hemiarthroplasty; SPAIRE; Direct Lateral Approach; Hip Surgery
MeSH Terms: conditions — Hip Fractures; Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct lateral approach (Active Comparator)
  Interventions: Procedure: Direct lateral approach
- Spaire approach (Experimental)
  Interventions: Procedure: SPAIRE

INTERVENTIONS:
Procedure: Direct lateral approach — The hip joint is approached from laterally, and parts of the gluteus medius tendon is released from the greater trochanter before the hip joint is entered from the anterior side.
  Other Names: Hardinge approach
  Arms: Direct lateral approach
Procedure: SPAIRE — The hip joint is entered from posterior, and the approach preserves the external rotators of the hip joint.
  Other Names: Muscle-sparing modification of the posterior approach
  Arms: Spaire approach

SUMMARY:
The HIFSAT study will compare the standard direct lateral approach to hemiarthroplasty to a new muscle sparing approach (SPAIRE) in femoral neck fracture patients.

DETAILED DESCRIPTION:
Femoral neck fractures are mostly treated with a hemiarthroplasty, where the fractured femoral head is replaced with a metal implant. The most common surgical approach to hemiarthroplasty has been the lateral approach, in which the gluteus medius tendon is partially released from the greater trochanter. Hip pain and limping is not uncommon after this approach has been used. A new surgical approach (SPAIRE) has been developed to alleviate this problem, and in this method the surgeon approaches the injured hip joint from posterior, preserving most of the muscles and tendons around the hip. This trial is designed to assess if this new SPAIRE approach leads to better results than the lateral approach in patients with femoral neck fractures.

ELIGIBILITY:
Inclusion Criteria:

* Femoral neck fracture
* Clinical indication for hemiarthroplasty
* Age over 50 years

Exclusion Criteria:

* Previous hip implants in the same hip
* Patients assessed to be in a terminal state with an expected survival of less than 1 week
* Other factors that makes follow-up impossible

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score ( HHS) | 4 months
  Harris Hip Score (HHS) is an outcome measure for hip-related symptoms. The score is based on both patient-reported information and clinical examination, and is administered by a qualified health care professional. It covers four domains: Pain, function, absence of deformity and range of motion. The score ranges from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Harris Hip Score (HHS) | 12 and 24 months
  Harris Hip Score (HHS) is an outcome measure for hip-related symptoms. The score is based on both patient-reported information and clinical examination, and is administered by a qualified health care professional. It covers four domains: Pain, function, presence of deformity and range of motion. The score ranges from 0 (worst) to 100 (best).
Oxford Hip score | 4,12 and 24 months
  Oxford Hip Score(OHS) is a patient reported outcome measure( PROM), OHS is designed to assess outcome after total hip replacement. It has 6 questions on pain and 6 questions on mobility. 5 categories of answer from worst to best. The range is 0-48.
EuroQol-5d-5l | 4,12 and 24 months
  EuroQol-5d-5l is a descriptive system comprises 5 dimensions: Mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the 5 dimensions can be combined into a 5-digit number that describes the patient's health state, and these digits can be converted into a single numerical value reflecting how the health state is according to the preferences of the general population of a country/region.
Trendelenburg test | 4,12 and 24 months
  This is a test to identify weakness in gluteal muscles, that can be seen in patients after hip surgery. Unilateral weakness in the gluteal muscles can for instance because nerve damage, trauma to the muscle or rupture of the tendon. The test will be performed as described by Hardcastle and Wade. The patient will be asked to raise their foot from the ground with 30º of hip flexion. The patient will be instructed to raise the non-stance side of the pelvis as high as possible with the examiner supporting the patient by holding their hands if needed. If the patient is not able to maintain this position for 30 seconds, or not being able to raise the hip of the non-stance side to above the level of the stance-side, the Trendelenburg test is considered positive.
New Mobility Score (NMS) | 4,12 and 24 months
  NMS consists of 3 questions about ambulation indoor, outdoor and the ability to go shopping. Each question has 4 alternative answers yielding 0-3 points, and the maximum score is 9.
Short Physical Performance Battery (SPPB) | 4, 12, an 24 months
  The Short Physical Performance Battery is an assessment tool made specific for screening of physical function among older adults. SPPB has 3 different tests: Balance, walking speed and rising from a chair. Scorings range from 0-12, best possible is 12.
Numerical Pain Rate Scale( NPRS) | 4, 12 and 24 months
  Unidimensional measure of pain intensity in adults, describing pain extreme from 0 no pain at all to 10 the worst pain imaginable.
Duration of surgery | 1.st day after surgery
  Duration of the operation in minutes
Preferred Walking Speed | 4,12 and 24 months
  A four-meter distance is marked on the floor, and the patients are instructed to walk this distance in their normal speed, as if they were walking down a street. The distance is walked twice, and the fastest speed is recorded. The subject can use any walking aids, and this is recorded.
Repeated Chair Stand Test | 4,12 and 24 months
  In the repeated chair stand test the participants are asked to fold their arms across their chest (the armrests shall not be not used) and stand up from the chair 5 times. This is timed by the examiner, and points are given from 0 to 4
Cumulated Ambulation Score | 1-5 days after surgery
  This will be recorded at day 1-3 for all patients. This score assesses the patients' early mobility by evaluating their ability to rise from bed, rise from a chair and walk indoor (walking aids permitted).
Timed up and go test | 4,12 and 24 months
  This test measures the time that the person uses to rise from a chair, walk three meters, turn around and walk back to the chair, and sit down again, turning 180 degrees. The person can use any mobility aids that he/she would normally use. The TUG test is being scored by the total time measured
Use of analgesia during admission | 1. day after surgery
  Analgesia during the first calendar day after surgery will be recorded as morphine equivalents according to a calculation table published by the Norwegian Directorate of Health.
Adverse events | 0-24 months
  Any adverse events will be recorded during the whole study period
Days Alive At Home (DAH) | 4,12 and 24 months
  Days alive and at home will be measured at 4,12 and 24 months. Patients wish to stay most of their lives at home, this measurement will tell us how long they could stay home and if they came home after their hip fracture.

OTHER OUTCOMES:
Grip strength | Day 1-5 after surgery, 4,12 and 24 months
  Sarcopenia is associated with low grip strength. The measurements will be taken with the patient sitting, with the elbow in 90° flexion and the shoulder adducted and neutrally rotated. The second handle position will be used for all participants. Two trials on each side will be conducted, starting with the dominant hand.
Patient Acceptable symptom State | 4,12 and 24 months
  Question about the patient´s satisfaction of the current state of their hip, and another question on whether they consider the treatment of their hip fracture to be a success or failure. They will also record a visual analogue scale of their satisfaction with the result of the surgery, ranging from "very satisfied" to "very dissatisfied".
Blood transfusion | 1st day after surgery until discharge, assessed up to 10 days
  Units of blood transfusion given to the patient during admission
Conventional radiographs of the operated hip | 1.st day after surgery and at 4 months after surgery
  Conventional radiographs will be taken postoperatively and at 4 months according to the standardized procedures for post-operative hip examinations of the radiology department. Using specialized computer software (Sectra Workstation IDS7 v.21 with orthopedic templating module Sectra Orthostation v15.1, Sectra AB, Linköping, Sweden), leg length difference, and hip offset compared to the uninjured hip will be recorded. In patients with a contralateral hip fracture this is not possible, but some of these patients will have available pre-fracture examinations that can be utilized for comparison. Femoral stem varus/valgus angulation (frontal view) and retroversion/anteversion (lateral view) will also be recorded
Body Mass Index | 4, 12 and 24 months
  Recorded with objective weight and height measurements.
Place of return from hospital | 4 months
  Place of return from hospital will be recorded, and at later visits the type of dwelling since the last visit will be recorded. We will differentiate between institution dwelling and community dwelling.
Clinical Frailty Scale | 4, 12 and 24 months
  Assessment of frail patients, grades from 1 (very fit patient) to 9 (terminally ill).

CONTACTS AND LOCATIONS:
Overall Officials: Siri Lillegraven, PhD, Study Chair — Diakonhjemmet Hospital
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway